CLINICAL TRIAL: NCT04666792
Title: PrEParing Family Planning Clinics to Streamline Integration of HIV Prevention Services for Young Women in Kenya
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Kenyatta National Hospital (Other Government); Kenya National AIDS & STI Control Programme (Other); Kisumu County Government (Unknown)
Responsible Party: Principal Investigator, Kenneth K Mugwanya, Assistant Professor, Global Health, School of Medicine and School of Public Health,, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00009583; R01MH123267 (NIH)
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: HIV Infections; Contraception; STI
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: This a programmatic stepped-Wedge cluster randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PrEP for HIV-1 uninfected for women accessing family planning (Other): Women accessing family planning will be assessed for HIV risk and PrEP eligibility. If eligible and willing to initiate PrEP, they will be provided PrEP in accordance with national guidelines as part of their standard of care at the family planning clinic.
  Interventions: Drug: PrEP

INTERVENTIONS:
Drug: PrEP — A fixed-dose, oral co-formulation of emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF) is the approved and preferred regimen for HIV-1 prevention in Kenya and the United States. The World Health Organization (WHO) recommends TDF-containing medications as PrEP, which includes TDF combined with FTC as well as potentially TDF alone and TDF combined with lamivudine (or 3TC, a medication closely related to FTC). Any TDF-containing medications that align with WHO and Kenya national guidelines for PrEP will be used. PrEP medication will come from clinic stocks.

SUMMARY:
This a prospective, open-label implementation project to catalyze integration of HIV prevention and PrEP care services for adolescent girls and young women in family planning clinics in Kenya.

DETAILED DESCRIPTION:
Investigators will conduct a stepped-wedge cluster-randomized programmatic project to integrate PrEP provision within a combination HIV prevention package in 12 family planning clinics in Kisumu, Kenya- a region with an HIV prevalence of up to 28% among young women. The project will optimize and sustain PrEP delivery with existing family planning staff, supported through training and ongoing technical assistance. The investigators will rigorously evaluate program reach, effectiveness, adoption, implementation, maintenance, and impact using validated implementation science frameworks and how clinics build new efficient delivery systems.

ELIGIBILITY:
Inclusion Criteria:

* Female of reproductive age
* Sexually active
* Able and willing to provide informed consent
* HIV negative, according to national HIV testing algorithm
* Has at least one risk factor for HIV as defined by the Kenya National AIDS and STI Control Program

Exclusion Criteria:

- Otherwise not eligible based on the above inclusion criteria

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25457 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of women accessing family planning services who are screened for HIV risk | up to 24 months
  Measure HIV risk screening completion among women receiving family planning services
Proportion of women accessing family planning services who uptake PrEP for HIV prevention | up to 24 months
  Measure PrEP initiation among women receiving family planning services

SECONDARY OUTCOMES:
PrEP adherence quantified by tenofovir drug levels in blood | up to 24 months
  Measure PrEP adherence among women who initiate PrEP
Proportion of women who remain HIV-negative | up to 24 months
  Assess HIV status of women receiving family planning services
Proportion of family planning clinics that implement PrEP provision | up to 36 months
  Measure number of clinics that provide PrEP
Proportion of targeted providers who are trained and provide PrEP | up to 24 months
  Measure number of providers in family planning clinics who implement PrEP
Proportion of core PrEP delivery components delivered per protocol | up to 24 months
  Measure fidelity to PrEP delivery procedures in family planning clinics
Facilitators and barriers to PrEP implementation | up to 24 months
  Mixed methods assessment of clinic readiness and ability to implement PrEP per protocol
Programmatic costs of providing PrEP in family planning clinics | up to 24 months
  Conduct micro-costing, cost-effectiveness, and budget impact analyses to estimate the programmatic costs of providing PrEP in family planning clinics
Develop data tools to expand and support delivery of family planning and HIV prevention services | up to 24 months
  Coordinate with key stakeholders to develop and refine data tools and clinical delivery products during project implementation

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Mugwanya, MBChB, MS, PhD, Principal Investigator — University of Washington
Locations (1):
- Kenyatta National Hospital, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mugwanya KK, Matemo D, Scoville CW, Beima-Sofie KM, Meisner A, Onyango D, Mugambi M, Feutz E, Grabow C, Barnabas R, Weiner B, Baeten JM, Kinuthia J; FP Plus Team. Integrating PrEP delivery in public health family planning clinics: a protocol for a pragmatic stepped wedge cluster randomized trial in Kenya. Implement Sci Commun. 2021 Dec 11;2(1):135. doi: 10.1186/s43058-021-00228-4. PMID 34895357